CLINICAL TRIAL: NCT01275989
Title: EAR ACUPUNCTURE EFFECTIVENESS IN REDUCING THE SIGNS AND SYMPTOMS OF STRESS AND ANXIETY
Acronym: EAEIRTSOSAA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Santander (Unknown)
Responsible Party: University São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 848/2009
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2010-06

CONDITIONS: Inclusion Criteria:; Voluntary Participation in the Study With Available Time for Submission to the Sessions, Which Occur Over Two Months.; Have a Score of Stress Medium, High or Very High in the LSS Questionnaire, Completion of the STAI and General Form.; Exclusion Criteria:; Pregnant Students.
MeSH Terms: interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 21 (Sham Comparator): sham acupuncture
  Interventions: Other: Ear acupuncture
- 15 (No Intervention): Control
  Interventions: Other: Ear acupuncture
- 20 (Active Comparator): intervention
  Interventions: Other: Ear acupuncture

INTERVENTIONS:
Other: Ear acupuncture

SUMMARY:
Randomized Controlled Trial found that levels of stress and anxiety of students ITIO, Ear and effective in reducing these levels. The LSS questionnaire and IDATE state were applied before, two months and two and a half months after the start of the applications, the STAI trait was applied once prior to the sessions. The sample comprised 56 individuals who had higher levels of stress above the average LSS 100 students who answered the questionnaires. Participants were divided randomly into three groups: control group with 15 patients without care, intervention group with 20 individuals using specific points for treatment and Group Sham at 21 points using individuals without indication for treatment of anxiety and stress. The results showed that the sham points decreased anxiety levels of participants.

DETAILED DESCRIPTION:
After checking the levels of stress and anxiety of students and workers from a school of massage and acupuncture concluded that auricular acupuncture in this study had significant results in reducing anxiety levels with the use of points and Ear Handle, but more studies are necessary so that it can be said that these points have sedating and calming effects for anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study with available time for submission to the sessions, which occur over two months.
* Have a score of stress medium, high or very high in the LSS questionnaire, completion of the STAI and general form.

Exclusion Criteria:

* Pregnant students. The only contraindication to this treatment is for pregnant women until the 3rd month of pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)